CLINICAL TRIAL: NCT04100161
Title: Skeletal Muscle Strain Injuries and the Connective Tissue: Optimal Nutritional Strategies During Rehabilitation After Acute Muscle Strain Injuries
Brief Title: Nutritional Strategies After Muscle Strain Injuries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Monika Lucia Bayer, Senior Researcher, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBH P147
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Muscle Strain, Multiple Sites
Keywords: muscle strain, atrophy, protein, rehabilitation
MeSH Terms: conditions — Sprains and Strains; Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein supplementation (Experimental): 20g protein supplementation twice daily for 3 months
  Interventions: Dietary Supplement: Protein supplementation; Procedure: Active rehabilitation
- Carbohydrate supplementation (Active Comparator): 20g maltodextrin supplementation twice daily for 3 months
  Interventions: Dietary Supplement: Carbohydrate supplementation; Procedure: Active rehabilitation

INTERVENTIONS:
Dietary Supplement: Protein supplementation — Daily dose of 40 g whey protein for 3 months
  Arms: Protein supplementation
Dietary Supplement: Carbohydrate supplementation — Daily dose of 40 g maltodextrin for 3 months
  Arms: Carbohydrate supplementation
Procedure: Active rehabilitation — Progressive rehabilitation following a muscle strain injury for 3 months

SUMMARY:
Muscle strain injuries are a particularly frequent type of sports injury in soccer, athletics, badminton/ tennis and cross-fit fitness, thereby affecting a broad range of popular leisure time activities. Depending on severity, sports-active individuals may experience long-term functional impairment and pain. Additionally, individuals having sustained one strain injury have a substantially increased risk of injuring the same muscle again. Strain injuries lead to long-term, potentially permanent, loss of muscle mass, thereby weakening the muscle. Muscle atrophy is likely a major factor in the high re-injury risk. Further, strain injuries are associated with a long-term inflammatory response.

In the current study, the investigators seek to study interventions to prevent the loss of muscle mass and elaborate on strategies to address the prolonged inflammation observed at the site of the injured muscle.

The primary aim of this study is to investigate the effect of protein supplementation on the reduction of muscle atrophy following a severe muscle strain injury in comparison to a carbohydrate supplement. As a second purpose, this study aims to elaborate on findings of prolonged inflammation intra-/ intermuscular by large-scale protein analysis and the characterization of cells active at the site of injury.

The study includes the following hypotheses:

1. Protein supplementation administered in combination with a gradually increasing loading regime (rehabilitation with weekly progression in load/ intensity) will be effective in reducing the injury-related loss of muscle mass.
2. The environment at the site of injury is not only pro-inflammatory, but contains proteins associated with proteolysis.
3. Cells belonging to the group of fibro-adipogenic progenitors will be accumulating intra- and inter-muscularly.

ELIGIBILITY:
Inclusion criteria:

* Sports-active men and women
* Acute muscle strain injury in either the calf muscles or the hamstring muscles
* Visible tear at the muscle-connective tissue interface visible on an US scan as a hypo-/ hyperechoic area

Exclusion criteria:

* Unwillingness to return to sports
* Claustrophobia
* Daily intake of non-steroidal anti-inflammatory drugs (NSAIDs) within 3 months prior to the strain injury
* Smoking
* Diagnosed or suspected type I or type II diabetes
* Diagnosed or suspected connective tissue and/or rheumatic diseases
* Any observed organ dysfunctions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Muscle volume | 3 months post injury
  Change in muscle volume in the injured muscle comparing immediate post injury scan with 3 months post scan plus comparison of change with healthy, contralateral muscle over the same time span.

SECONDARY OUTCOMES:
Muscle volume | 12 months post injury
  Change in muscle volume in the injured muscle comparing immediate post injury scan with 12 months post scan plus comparison of change with healthy, contralateral muscle over the same time span.
Isokinetic muscle strength | 3 months post injury
  Change in muscle strength in the injured leg compared to muscle strength in healthy, contralateral muscle
Isokinetic muscle strength | 6 months post injury
  Change in muscle strength in the injured leg compared to muscle strength in healthy, contralateral muscle
Isokinetic muscle strength | 12 months post injury
  Change in muscle strength in the injured leg compared to muscle strength in healthy, contralateral muscle
Fat infiltration | 3 months post injury
  Assessment of fat content in the injured muscle comparing immediate post injury scan with 3 months post scan plus comparison of change with healthy, contralateral muscle over same time range
Fat infiltration | 12 months post injury
  Assessment of fat content in the injured muscle comparing immediate post injury scan with 12 months post scan plus comparison of change with healthy, contralateral muscle over same time range
Injury screening Questionnaire | 3 months post
  Assessment of subjective symptoms and pain during sports and daily activities
Injury screening Questionnaire | 6 months post
  Assessment of subjective symptoms and pain during sports and daily activities
Injury screening Questionnaire | 12 months post
  Assessment of subjective symptoms and pain during sports and daily activities
Ultrasound images | Baseline (Acute post injury)
  Fascicle length measurement, pennation angle, mechanical properties of the muscle (- tendon unit) in the injured and healthy, contralateral muscle
Ultrasound images | 3 months post injury
  Fascicle length measurement, pennation angle, mechanical properties of the muscle (- tendon unit) in the injured and healthy, contralateral muscle
Ultrasound images | 6 months post injury
  Fascicle length measurement, pennation angle, mechanical properties of the muscle (- tendon unit) in injured and healthy, contralateral muscle
Ultrasound images | 12 months post injury
  Fascicle length measurement, pennation angle, mechanical properties of the muscle (- tendon unit) in the injured and healthy, contralateral muscle
Assessment injury exudate | Within 7 days post injury
  Assessment and characterization of cells and soluble factors released after a strain injury into the intra-/ intermuscular space
Assessment injury exudate | <1 week post injury -12 weeks post injury
  Assessment and characterization of cells and soluble factors released after a strain injury into the intra-/ intermuscular space

CONTACTS AND LOCATIONS:
Overall Officials: Monika L Bayer, PhD, Principal Investigator — Institute of Sports Medicine, Copenhagen
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Nielsine Nielsen Vej 11, Building 8, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual de-identified participant data or other documents such as study protocol will not be shared with any third party. A potential change in the data sharing plan after registration will be acknowledged as a statement in a submitted/ published manuscript. A change in the data sharing statement will furthermore be updated in the registry record.

REFERENCES:
- [Derived] Mertz KH, Sorensen HH, Lorentz C, Johansen E, Fredskild NU, Wulff MW, Svensson RB, Kjaer MB, Linden FH, Kjaer M, Bayer ML. Effects of Protein Supplementation During Early Rehabilitation on Muscle Volume and Function After Acute Muscle Strain Injuries: A Randomized Controlled Trial. Scand J Med Sci Sports. 2025 Apr;35(4):e70043. doi: 10.1111/sms.70043. PMID 40145631